CLINICAL TRIAL: NCT02020655
Title: Measurement of Cytokines (IL-1α) After Shear- Force Application at the Skin
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL46877.068.13
Record Dates: First submitted 2013-11-05; First posted 2013-12-25 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Pressure Ulcers, Bedsores, Decubitus Ulcer
Keywords: IL-1 alpha, Sebutape, shear- force
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 10 healthy volunteers: Shear- force model
  Interventions: Other: Shear- force model

INTERVENTIONS:
Other: Shear- force model — Shear- force model

SUMMARY:
Background: A pressure ulcer is localized tissue injury to the superficial layer of the skin and/ or the underlying tissue. Pressure ulcers are most likely to develop in skin areas exposed to pressure, shear and friction. Shear- force is an important contributing factor and wound dressing are possibly capable to reduce shear force at the skin. At this moment there's no good marker to detect the effect of shear- force at the skin. A potential marker could be cytokines (IL-1α) which are released after mechanical loading of the skin. A previous study have shown a significant increased level of IL-1α after the application of pressure. We want to investigate if these cytokines are significant increased after the application of shear- force at the skin.

Objective: The objective of this study is to gather knowledge about cytokine concentrations (IL-1 α) in the skin of healthy volunteers after the application of shear- force. We want to use this knowledge in the future to investigate if different prophylactic wound dressings are capable to reduce shear force at the skin. This could be interesting in the prevention of pressure ulcers.

Study design: With the use of a special developed shear- force model are we going to administer 20 Newton (2 kg) shear at the palmar side of the under arm in 10 healthy volunteers for 30 minutes. As a control we ware going to put the shear- force model at the other arm without the application of shear- force. Before the use of the shear- force model we will perform cytokine measurements with the use of Sebutape. Sebutape is capable to absorb cytokines from the skin. After the use of the shear force- model we will perform cytokine measurements again. Then we will extract the cytokines from the Sebutape with the use of ELISA.

Study population: 10 Healthy volunteers Age 18- 30 years

Primary outcome: IL-1 α concentration (pg/ml)

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 30 years
* BMI 20 -30
* Braden score > 20

Exclusion Criteria:

* Trauma arms
* Skin diseases (eczema, psoriasis)
* Inability to give informed consent
* Muscle disorders
* malignancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
IL-1 α concentration (pg/ml) | up to 24 hours
  With the use of a special developed shear- force model are we going to administer 20 Newton (2 kg) shear at the palmar side of the under arm in 10 healthy volunteers for 30 minutes. As a control we ware going to put the shear- force model at the other arm without the application of shear- force. Before the use of the shear- force model we will perform cytokine measurements with the use of Sebutape. Sebutape is capable to absorb cytokines from the skin. After the use of the shear force- model we will perform cytokine measurements again.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, MD, PhD, Study Chair — Department of surgery, Maastricht University Medical Centre
Locations (1):
- Maastricht University medical Centre, Maastricht, Limburg, Netherlands